CLINICAL TRIAL: NCT04092335
Title: Evaluation of Adam's Forward Bend Test and Smartphone Application in Screening of Adolescent Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Karima Abdelaty Hassan, Lecturer, Cairo University
Other Study IDs: P.T.REC/012/002051
Record Dates: First submitted 2019-09-14; First posted 2019-09-17 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Scoliosis is a lateral curvature of the spine when the Cobb´s angle more than 10˚ on the frontal plane. Curve detection before skeletal maturation gives a good opportunity for early treatment or prevention of curve progression. Purpose of this study was to evaluate Adam's Forward Bend Test and Scoliometer HD in screening of Adolescent Idiopathic Scoliosis

DETAILED DESCRIPTION:
The student was asked to stand erect, knees straight, feet at the same level and hands freely hanging.

They was observed from the back for shoulders, pelvic, and knees level. Student was asked to bend forward with his knees straight, feet together and hands freely and loosely hanged(Forward Bend Test).

Scoliosis was detected with rib cage rotation and hump appearance (positive test).

Absence of hump appearance means negative test. After Forward Bend, the students were screened using the Scoliometer HD Application.

The students were asked to bend forward with arms dangling and palms pressed together. The smart phone (Scoliometer HD) was placed on the student back with the central dark area in the application placed on the spinous processes of the lumber and thoracic regions to measure the angle of trunk rotation. Students with a scoliometer HD reading ≥7 degrees (≥20 ̊ Cobb's angle) were referred to orthopedic consultation and their parents were informed about the findings of the screening by the school manager and social worker.

Then the data were collected for statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* Age range from 10 to 15 year.
* Males ( parents of girls refused their participation).
* Students who have structural scoliosis.

Exclusion Criteria:

* Congenital deformities.
* Neuromuscular disorder (Cerebral palsy and spinal muscle atrophy).
* Syndromic disorders (Muscular dystrophy, Osteogenesis imperfect and spinabifida).

Ages: 10 Years to 15 Years | Sex: Male
Age Groups: Child
Study Population: Male students with age range 10-15 years
Sampling Method: Non-Probability Sample
Enrollment: 840 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Appearance of hump measured by Forward Bend Test | 20 minutes
  Students were asked to bend forward with his knees straight, feet together and hands freely and loosely hanged. Scoliosis were detected with rib cage rotation and hump appearance (positive test). Absence of hump appearance means negative test.
Angle of trunk rotation (ATR) measured by Scoliometer HD application | 20 minutes
  The students were asked to bend forward with arms dangling and palms pressed together. The smart phone (Scoliometer HD) was placed on the student back with the central dark area in the application placed on the spinous processes of the lumber and thoracic regions to measure the angle of trunk rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Nasr A. Abdelkader, PhD, Principal Investigator — Lecturer,Cairo University
Locations (1):
- Cairo university, Giza, Egypt